CLINICAL TRIAL: NCT01356017
Title: A Randomized, Open-label, Multiple Doses, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction and Safety of Telmisartan Between Free Combination of Telmisartan and S-amlodipine and Telmisartan Monotherapy in Healthy Male Volunteers
Brief Title: CKD-828 Drug Interaction Study (Telmisartan)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Jin Kim/ Director, Clinical Research Department
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 130HPS11C
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — Telmisartan; levamlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Free combination of Telmisartan and S-amlodipine (Experimental): Subjects received Telmisartan 80mg and S-amlodipine 5mg once a day for 9 days. And subjects doesn't take any medications for 19 days.
  Interventions: Drug: Telmisartan 80mg, S-amlodipine 5mg
- Telmisartan monotherapy (Active Comparator): Subjects received Telmisartan 80mg once a day for 9 days. And subjects doesn't take any medications for 19 days.
  Interventions: Drug: Telmisartan 80mg

INTERVENTIONS:
Drug: Telmisartan 80mg, S-amlodipine 5mg — Telmisartan 80mg and S-amlodipine 5mg, Oral, Once a day, for 9 days + Wash out (19 days)
  Other Names: Micardis 80mg, Anydipine S 5mg
  Arms: Free combination of Telmisartan and S-amlodipine
Drug: Telmisartan 80mg — Telmisartan 80mg, Oral, Once a day, for 9 days + Wash out (19 days)
  Other Names: Micardis 80mg
  Arms: Telmisartan monotherapy

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetic drug interaction and safety of Telmisartan between free combination of Telmisartan and S-amlodipine and Telmisartan monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 50 aged in healthy males
* Weight more than 55kg, BMI 19kg/m2-26kg/m2 at the period of screening
* 100mmHg ≤ sit SBP < 140mmHg and 60mmHg ≤ sit DBP < 90mmHg and 50 per/min ≤ Pulse rate < 95 per/min
* AST, ALT, Total bilirubin < UNL x 1.5
* Signed the informed consent from prior to the study participation

Exclusion Criteria:

* Have history of significant hepatic, renal, gastrointestinal, pulmonary, musculoskeletal, endocrine, neuropsychiatric, hematologic, cardiovascular diseases
* Have a gastrointestinal disease(ex : Crohn's disease, gastrointestinal ulcer) or surgery(except for Appendectomy, hernia repair) affected by the absorption of medications
* galactose intolerance or Lapp lactase deficiency or glucose-galactose malabsorption
* Hypersensitivity reactions to drugs or clinically significant hypersensitivity reactions in the history of telmisartan or Amlodipine
* drug abuse, or have a history of drug abuse showed a positive for the Triage TOX drug on urine : amphetamine, barbiturate, cocaine, opiates, benzodiazepines, THC(cannabinoids), methadone etc.
* Subject takes herbal medicine within 30 days, ethical drug within 14 days, OTC within 7 days before the beginning of study treatment
* unusual diet affected by the absorption, distribution, metabolism, excretion of medications
* Subject who treated with any investigational drugs within 90 days before the beginning of study treatment
* Previously donate whole blood within 60 days or component blood within 30 days or transfusion within 30 days
* Subject who takes inhibitors and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30 days
* A heavy caffeine consumer (caffeine > 5 units/day),
* A heavy alcohol consumer (alcohol > 21 units/week, 1 unit=pure alcohol 10mL) or cannot stop drinking
* A heavy smoker (cigarette > 20 cigarettes per day)
* Positive for Hepatitis B, Hepatitis C, HIV or syphilis
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result, EKG result

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Telmisartan AUC | 0, 192, 192.5, 193, 193.5, 194, 195, 196, 197, 198, 200, 202, 204, 216 hr

SECONDARY OUTCOMES:
Telmisartan Cmax | 0, 192, 192.5, 193, 193.5, 194, 195, 196, 197, 198, 200, 202, 204, 216 hr
Telmisartan Tmax | 0, 192, 192.5, 193, 193.5, 194, 195, 196, 197, 198, 200, 202, 204, 216 hr

CONTACTS AND LOCATIONS:
Overall Officials: Kyun S Bae, Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Noh YH, Lim HS, Kim MJ, Kim YH, Choi HY, Sung HR, Jin SJ, Lim J, Bae KS. Pharmacokinetic interaction of telmisartan with s-amlodipine: an open-label, two-period crossover study in healthy Korean male volunteers. Clin Ther. 2012 Jul;34(7):1625-35. doi: 10.1016/j.clinthera.2012.05.010. Epub 2012 Jun 19. PMID 22721873